CLINICAL TRIAL: NCT05937776
Title: Development of Activity MRI (aMRI): Direct Comparison to PET in Human Subjects
Brief Title: Developing a New Metabolic Imaging Approach (aMRI) for Evaluating Neurological Disease in Patients With Gliomas
Status: Recruiting | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Martin Pike, Ph.D., Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: STUDY00024504; NCI-2023-04867 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Fluorodeoxyglucose F18; Fluorine-18; gadoterate meglumine; gadolinium 1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetraacetate; Magnetic Resonance Spectroscopy; Contrast Media; X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic (¹⁸FDG PET, MRI): Patients receive ¹⁸FDG IV, then 60 minutes later undergo simultaneous MRI and PET scanning. During this scanning period, patients will receive gadoterate meglumine IV to obtain post-contrast MRI. Total scanning time will take 45-60 minutes.
  Interventions: Other: Fludeoxyglucose F-18; Other: Gadoterate Meglumine; Procedure: Contrast-enhanced Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: ¹⁸FDG; 2-Deoxy-2-(18F)Fluoro-D-Glucose; 2-F18-Fluoro-2-deoxy-D-glucose; Fludeoxyglucose (18F); 105851-17-0; 2-F18-Fluoro-2-deoxyglucose; FDG; fludeoxyglucose F 18; Fluorine-18; Fludeoxyglucose F18; 2-Fluoro-2-deoxy-D-Glucose
Other: Gadoterate Meglumine — Given IV
  Other Names: 92943-93-6; DOTAREM; Gd-DOTA
Procedure: Contrast-enhanced Magnetic Resonance Imaging — Undergo PET/contrast-enhanced MRI
  Other Names: CONTRAST ENHANCED MRI; Contrast-enhanced MRI; MRI With Contrast
Procedure: Positron Emission Tomography — Undergo PET/contrast-enhanced MRI
  Other Names: Medical Imaging; PET; PET Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This is an observational study to compare the utility of the novel aMRI approach in human brain to the standard of care imaging approach for diagnosing and assessing glioma. Tumor cells have altered metabolism compared to normal cells.This makes metabolic activity imaging useful for diagnosing and assessing neurological disease. However, current options for metabolic activity imaging are limited. Metabolic activity imaging is primarily conducted using positron emission tomography (PET) with a radioactive tracer called fludeoxyglucose F-18 (¹⁸FDG). A PET scan is a procedure in which a small amount of radioactive glucose (¹⁸FDG) is injected into a vein, and a scanner is used to make detailed, computerized pictures of areas inside the body where the glucose is taken up. PET imaging is very expensive and is usually much less available than other imaging techniques such as magnetic resonance imaging (MRI). MRI uses radiofrequency waves and a strong magnetic field to provide clear and detailed pictures of internal organs and tissues. While MRI is more available than PET, it isn't as useful in evaluating metabolic activity. Unlike standard MRI, the aMRI approach uses new ways of analyzing MRI images that provides information about tumor cell metabolic activity. Via direct comparison with a standard metabolic imaging approach, ¹⁸FDG PET, this clinical trial will assess the validity of aMRI as a metabolic imaging approach for evaluating neurological disease in patients with glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Characterize how the metabolic aMRI parameter kᵢₒ*V differs in tumor versus (vs) normal brain. Researchers will assess the validity of aMRI as a metabolic imaging approach via direct comparison with a standard metabolic imaging approach, ¹⁸FDG PET.

SECONDARY OBJECTIVES:

I. Post-gadolinium (Gd) T1 MRI will be used to distinguish the contrast-enhancing "ring" region indicating the metabolically active tumor periphery from the less viable and/or necrotic tumor core. The utility of aMRI to differentially assess the metabolically active tumor periphery and necrotic core regions will be determined and compared to that of ¹⁸FDG PET (SUVmax).

II. Characterize how the metabolic aMRI parameter kᵢₒ*V differs in the various normal appearing brain sub-regions unaffected by tumor, in comparison to ¹⁸FDG PET.

EXPLORATORY OBJECTIVE:

I. To compare how the aMRI metabolic parameter kᵢₒ*V within disease lesions change with different disease types, their disease stage, and their treatment status.

OUTLINE:

Patients receive ¹⁸FDG IV, then 60 minutes later undergo simultaneous MRI and PET scanning. During this scanning period, patients will receive gadoterate meglumine IV to obtain post-contrast MRI. Total scanning time will take 45-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 18 years of age) with glioma who require MRI and ¹⁸FDG-PET imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with glioma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean values of kᵢₒ*V of the entire tumor region | Up to 1 year
  In subjects with glioma brain tumors, outlines of tumor regions will be defined by post-contrast T1 magnetic resonance images. Mean values of kᵢₒ*V of the entire tumor region will be obtained and in normal-appearing contralateral regions for comparison. The profile of mean values in these regions will be evaluated for efficacy in metabolically distinguishing them, and evaluated for correlation with the co-registered flurodeoxyglucose F-18 (¹⁸FDG) positron emission tomography (PET) (standardized uptake value maximum [SUVmax]) data. The observation of robust correlation with PET, would validate activity magnetic resonance imaging (aMRI) as a metabolic sensor.

SECONDARY OUTCOMES:
Mean value of kᵢₒ*V in the tumor periphery and core regions | Up to 1 year
  Mean values of kᵢₒ*V will be obtained in the tumor periphery and core regions. The data will be evaluated for utility in metabolically distinguishing them, and evaluated for correlation with the co-registered ¹⁸FDG PET (SUVmax) data.
kᵢₒ*V in different normal appearing brain sub-regions, unaffected by tumor | Up to 1 year
  Will quantify the aMRI metabolic parameter kᵢₒ*V in different normal appearing brain sub-regions, unaffected by tumor, as defined by registration to a human brain Atlas. The profile of mean values in these regions will be evaluated for efficacy in metabolically distinguishing them, and evaluated for correlation with the simultaneously obtained and co-registered ¹⁸FDG PET (SUVmax) data.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pike, Ph.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States